CLINICAL TRIAL: NCT04576273
Title: Enterobius Vermicularis in Appendectomy Specimens; Clinicopathological Assessment
Brief Title: Enterobius Vermicularis Infestation of the Appendix
Status: Completed | Type: Observational
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Aabdulkarim Hasan, Lab Director, Al-Azhar University
Other Study IDs: 3003
Record Dates: First submitted 2020-09-23; First posted 2020-10-06 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-09

CONDITIONS: Parasitic Disease
MeSH Terms: conditions — Parasitic Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-parasitic
  Interventions: Diagnostic Test: Pathology examination
- Parasitic
  Interventions: Diagnostic Test: Pathology examination

INTERVENTIONS:
Diagnostic Test: Pathology examination — Gross and microscopic evaluation

SUMMARY:
This study identifies the incidence of appendiceal Enterobius vermicularis (E.v) infestation in all the patients undergoing appendectomy and evaluates the relationship between E.v infestation of the appendix and the acute appendicitis.

DETAILED DESCRIPTION:
All the patients undergoing appendectomy surgical procedure for clinical picture of acute appendicitis in 3-years period at our referral hospital were evaluated to pick up the Enterobius vermicularis infestation of the appendix. These cases were evaluated for clinico-laboratory characterization to define the incidence in our country and the relationship between the E.v and initiation of the the inflammatory process to study the possibility of limitation of surgical intervention in acute abdomen conditions.

ELIGIBILITY:
Inclusion Criteria:

All routine examined appendectomy specimens

Exclusion Criteria:

Cases with clinical suspicion of tumor Cases attached to the colectomy specimens

Ages: 4 Years to 90 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Saudi and non- Saudi patients suffering from acute appendicitis symptoms
Sampling Method: Non-Probability Sample
Enrollment: 1150 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Association between acute inflammation and Enterobius vermicularis infestation | 3 years
  All the studied Enterobius vermicularis cases will be evaluated microscopically to record the count of acute inflammatory cells per millimeter (mm) and per High Power Field (HPF) using the microscope scale measurement. This count will be compared with the inflamed appendectomy specimens without Enterobius infestation to assess the hypothesis of the association between the Enterobius infestation and the acute appendicitis. Also special stain (congo red) will be implicated in some indicated cases to detect eosinophils, eosinophils will be positively staines (orange color stain means positive) if the stain is faint that means negative and the cell is not eosinophil
Incidence of Appendiceal Enterobius vermicularis | 3 years
  An incidence of Enterobius infestation will be assessed by studying all the received specimens during a 3 years-period using formatting a master sheet and processing in Excel program

CONTACTS AND LOCATIONS:
Locations (1):
- Abdulkarim Hasan, Baljurashi, Saudi Arabia